CLINICAL TRIAL: NCT01995539
Title: Use of iPro™2 in Real Life Diabetes Management of Type 2 Patients in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP274
Record Dates: First submitted 2013-11-08; First posted 2013-11-26 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iPro2 Use (Experimental): All subjects wearing iPro2, having therapy regimens, and having baseline and EOS A1C tests
  Interventions: Behavioral: therapy regimen

INTERVENTIONS:
Behavioral: therapy regimen — Subjects will be recommend changes in therapy regimens.

SUMMARY:
The purpose of the India iPro2 study is to demonstrate that iPro2 Continuous Glucose Monitoring System (CGMS) evaluation enables Health Care Professional (HCP)s treating patients in India with type 2 diabetes to get a better understanding of their patient's metabolic fluctuations, and support appropriate therapeutic intervention.

DETAILED DESCRIPTION:
The study will be designed to demonstrate the value of iPro2 in real-world diabetes management in type 2 patients in India. It will be an interventional post-market, prospective, multi-center study with a data review performed after 30 subjects have completed the trial.

During the course of the study, patients will undergo two iPro2 evaluations:

* First iPro2 test (Visit 1 [application] & 2 [removal])
* Second iPro2 test (Visit 3 [application] & 4 [removal])

Patient and HCP questionnaires will be administered at Visit 1, 2, 3, 4 and 5. These questionnaires aim to assess the impact of an iPro2 evaluation on the physicians understanding of their patient's metabolic fluctuations and its support of therapeutic interventions. They will also investigate the subjects understanding (both pre & post iPro2 evaluation) of the concept of glycemic variability and the importance of compliance to HCP recommendations.

ELIGIBILITY:
Inclusion criteria:

1. Subject is > 18 years to ≤ 70 years of age
2. Subject has been diagnosed with type 2 diabetes mellitus for at least 1 year and is currently being treated with an oral anti-hyperglycemic medication and/or insulin
3. Subject's A1C > 8.0% to ≤ 10% conducted in the last 4 weeks
4. Subject, or legal representative, has signed the study Patient Informed Consent Form (PIC)
5. Subject is willing to comply with the study procedures

Exclusion criteria:

1. Subject is unable to tolerate tape adhesive in the area of sensor placement
2. Subject is pregnant, or is expecting to become pregnant during the course of the trial per Investigator discretion.
3. Subject has no experience with SMBG and blood glucose meter use
4. Subject has undergone an iPro evaluation during the past 6 months
5. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, rash, Staphylococcus infection)
6. Subject is actively participating or planning to actively participate in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
7. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
8. Subject has unresolved alcohol or drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jothydev Kesavadev, MD, Principal Investigator — Jothydev's Diabetes and Research Centre; Mohan V, MD, Principal Investigator — Madras Diabetes Research Foundation; Vijay Viswanathan, MD, Principal Investigator — M.V Hospital for Diabetes Research centre; Ambrish Mithal, MD, Principal Investigator — Medanta Institute of Clinical Research; Manoj Chawla, MD, Principal Investigator — Lina Diabetes Care Mumbai Diabetes Research Centre; Rajiv Kovil, MD, Principal Investigator — Dr.Kovil's Diabetes Care centre; Banshi Saboo, MD, Principal Investigator — DIA Care; Sunil Jain, MD, Principal Investigator — TOTALL Diabetes Hormone Institute; Abhay Mutha, MD, Principal Investigator — Diabetes Care & Research Center; Shehla Shaikh, MD, Principal Investigator — K.G.N DIABETES AND ENDOCRINE CENTRE; Dharmen Punatar, MD, Principal Investigator — Diab Care Centre; Scott Lee, MD, Study Director — Medtronic Diabetes
Locations (11):
- India (11):
  - Madras Diabetes Research Foundation, Gopālapuram, Chennai
  - DIA Care, Ahmedabad, Gujarat
  - Medanta, Gurgaon, Haryana
  - Jothydev's Diabetes and Research Centre, Trivandrum, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - K.G.N Diabetes and Endocrine Centre, Mumbai, Maharashtra
  - Lina Diabetes Care Centre, Mumbai, Maharashtra
  - Dr.Kovil's Diabetes Care centre, Mumbai, Maharashtra
  - Diab Care Center, Mumbai, Maharashtra
  - Diabetes Care & Research Center, Pune, Maharashtra
  - M.V Hospital for Diabetes Research centre, Chennai, Tamil Nadu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iPro2 Use
Started | 181
Completed | 148
Not Completed | 33
Not completed — Screening Failure | 1
Not completed — Withdrawal by Investigator | 15
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 5
Not completed — Subject missed visit 3,4, came in for V5 | 1

BASELINE CHARACTERISTICS:
Arm/Group | iPro2 Use
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 111
Region of Enrollment [Number; unit: participants]
  India | 181

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at 3 Months
Description: Descriptive analysis of change in A1C from baseline to end of 3-month study period
Time Frame: 3 months
Population: 181 subjects consented and screened; 1 subject screen failed; 148 subjects completed study; 32 subjects not completed study.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | iPro2 Use
Number analyzed (Participants) | 148
percent | -0.6 (1.11)

2. Secondary Outcome: Number of Serious Adverse Device Effects (SADE).
Description: Evaluation of incidence of SADE during the study.
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | iPro2 Use
Number analyzed (Participants) | 181
events | 0

ADVERSE EVENTS:
Time Frame: 3 Month
Arm/Group | iPro2 Use
All-Cause Mortality (participants affected / at risk) | 0/181
Serious Adverse Events (participants affected / at risk) | 0/181
Other Adverse Events (participants affected / at risk) | 5/181
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iPro2 Use (N=181)
Pricking sensation at insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
BLEEDING AT SENSOR INSERTION SITE (General disorders) | 1 (1)
itching at sensor insertion site (Skin and subcutaneous tissue disorders) | 2 (2)
Pain at insertion site area (General disorders) | 2 (2)
Skin irritation at sensor insertion site (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days